CLINICAL TRIAL: NCT01964417
Title: The Comparative Study Between Bowel Preparation Method: 4L-split Dose of PEG Solution, Low-volume PEG Plus Ascorbic Acid Focusing on the Bowel Cleansing Efficacy, Patients' Affinity to Preparation Solution and Mucosal Injury
Brief Title: The Comparative Study Between Bowel Preparation Method
Acronym: CSBPM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jongha Park, Inje University, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PEG-0488
Record Dates: First submitted 2013-09-30; First posted 2013-10-17 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Colonoscopy
Keywords: BOWEL PREPARATION; PEG; Low-volume PEG Plus Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4L-split Dose of PEG Solution (Active Comparator): 4L-split Dose of PEG Solution for bowel preparation
  Interventions: Drug: Colonoscopy after bowel cleansing
- Low-volume PEG Plus Ascorbic Acid (Active Comparator): Low-volume PEG Plus Ascorbic Acid for bowel preparation
  Interventions: Drug: Colonoscopy after bowel cleansing

INTERVENTIONS:
Drug: Colonoscopy after bowel cleansing

SUMMARY:
The purpose of this study is to compare the efficacy, acceptability and preparation-induced mucosal inflammation of PEG + ascorbic acid vs. PEG for colonoscopy.

DETAILED DESCRIPTION:
This was a prospective randomized single-blinded clinical trial of ambulatory patients to assess the efficacy of bowel preparation and preparation-induced mucosal inflammation.

Endoscopists who were blinded to the preparation taken, assessed both bowel cleansing by using the Ottawa bowel preparation assessment tool and preparation-induced mucosal inflammation. Acceptability was assessed by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who want colonoscopy purposing screening among adults between the age of 20~65

Exclusion Criteria:

* Under the age of 20, older than 65, pregnant or lactating women, intestinal obstruction, structural intestinal disease, hypothyroidism, gastrointestinal motility, renal failure, congestive heart failure, liver failure, electrolyte abnormalities, who refused research informed consent, inflammatory bowel disease, the obvious symptoms of the disease in patients with lower gastrointestinal (bloody stools, diarrhea, etc.)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison of colon cleansing between the two solutions using Ottawa scale | 3month

CONTACTS AND LOCATIONS:
Overall Officials: Jongha Park, MD, Principal Investigator — Inje University
Locations (1):
- Haeundae Paik Hospital, Busan, South Korea